CLINICAL TRIAL: NCT06135376
Title: E-PAUse: Encouraging Proper Antibiotic Use in Outpatient Setting
Acronym: E-PAUse
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hamad Medical Corporation (Industry)
Collaborators: Primary Health Care Corporation, Qatar (Other Government)
Responsible Party: Principal Investigator, Adeel Ajwad Butt, Senior Consultant in Infectious Disease, Hamad Medical Corporation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MRC-01-23-076
Record Dates: First submitted 2023-11-09; First posted 2023-11-18 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Drug Use
Keywords: Prescription rate; Antibiotics;

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control groups with single intervention (Active Comparator): The control groups will each receive a single intervention which will be selected at random.
  Interventions: Behavioral: comprehensive multi-component interventions
- Experimental group with 4 interventions (Experimental): 2 Primary Health Care Centers (PHCCs) will receive the comprehensive multi-component intervention, which consists of four elements:
  1. Option for deferred prescription fulfilment.
  2. Education of staff regarding appropriate uses of antibiotics.
  3. algorithm-driven decision support tool.
  4. Feedback on individual and group performance. The training will be repeated at monthly intervals over the 6-month intervention period.
  Interventions: Behavioral: comprehensive multi-component interventions

INTERVENTIONS:
Behavioral: comprehensive multi-component interventions — It is a combination of educational and behavioral interventions. 4 PHCCs will be randomized to 2 groups: 2 PHCCs will receive single intervention and 2 PHCCs will receive all 4 interventions.

SUMMARY:
Specific Aim 1: To determine the knowledge, attitude, and practice (KAP) of PHCC physicians regarding appropriate prescription of antibiotics in the outpatient setting.

Hypothesis 1a: PHCC physicians will have adequate theoretical knowledge regarding use of antibiotics for upper respiratory tract infections.

Hypothesis 1b: Despite adequate theoretical knowledge, fear of complications of untreated infection and patient demand and expectations will drive inappropriate antibiotic prescription for upper respiratory tract infections

Specific Aim 2: To test the effectiveness of a comprehensive multi-component intervention in a cluster randomized trial upon rate of antibiotics prescription for upper respiratory tract infections in individuals aged > 2 years presenting to primary care by PHCC physicians Hypothesis 2: Compared with a single intervention, a comprehensive multi-component intervention package will be associated with a significant reduction in inappropriate antibiotic prescription.

Investigators will conduct this study in the Primary Healthcare Center (PHCC) setting in Qatar. Investigators will identify four large PHCCs from the existing active centers. The study has 2 parts. Part 1 corresponds to specific aim 1 and comprises of a KAP survey which will be carried out in all four PHCCs and will include all physicians. Part 2 corresponds to specific aim 2 and is a cluster randomized clinical trial in which Investigators will randomize the four PHCCs into two groups.

First group (2 PHCCs) will receive training in appropriate documentation of infections and antibiotics prescription and will continue to provide usual care. Second group (2 PHCCs) will receive the comprehensive multi-component intervention, which consists of four elements:

1. Option for deferred prescription fulfilment;
2. Education of staff regarding appropriate uses of antibiotics,
3. algorithm-driven decision support tool,
4. Feedback on individual and group performance.

DETAILED DESCRIPTION:
As above.

ELIGIBILITY:
Inclusion Criteria:

* Patients >2 years old presenting to any of the selected PHCCs (rationale: signs and symptoms of bacterial infection in very young children are more non-specific and empiric antibiotics are often indicated due to serious consequences of unrecognized and untreated bacterial infections)
* Presenting with acute (<1 week of symptoms) upper respiratory tract infection (URTI) like illness including

  * common cold/acute rhinitis/nasopharyngitis
  * laryngitis/laryngotracheitis
  * Acute bronchitis
  * acute otitis media
  * influenza (confirmed or influenza-like illness)
  * pharyngitis/tonsillitis
  * acute sinusitis

Exclusion Criteria:

* Known immune compromised status, e.g., cystic fibrosis, cancer, organ transplant recipient.
* On immune suppressive therapy for any duration (e.g., steroids, disease modifying antirheumatic agents; cancer chemotherapy, anti-rejection drugs, etc.) in one year prior to presentation
* Known or diagnosed bacterial cause of infection.
* Severe systemic illness requiring referral to the emergency department or hospitalization within 24 hours of presentation
* Known or suspected chronic obstructive pulmonary disease. Asplenic patients (anatomic or functional)

Ages: 2 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100000 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Total number of antibiotics courses prescribed for URTIs | Primary Analysis 11 months; Final analysis 24 months
  For each recorded diagnosis of URTI, investigators will count the number of persons who received an antibiotic prescription. All prescriptions regardless of drug, dose, route of administration and duration will be counted. Only one prescription per 30-day period will be counted to exclude those with ongoing, evolving, or unresolved infection.
Proportion of antibiotics prescription dispensed for an inappropriate use | Total 11 months for primary analysis; Follow-up up to 36 months
  For each antibiotic prescription written for a URTI diagnosis, investigators will determine the appropriateness of antibiotics based on our previously published criteria.

SECONDARY OUTCOMES:
Rates of hospitalization in 28 days after the PHCC visit | Total 11 months for primary analysis; Follow-up up to 36 months
  Number of hospitalizations within 28 days of the index visit
Rates of ED visits in 28 days after the PHCC visit | Total 11 months for primary analysis;
  Number of ED visits within 28 days of the index visit

CONTACTS AND LOCATIONS:
Overall Officials: Adeel A. Butt, MBBS, MS, Principal Investigator — Hamad Medical Corporation
Locations (1):
- PHCC, Doha, Qatar

REFERENCES:
- [Derived] Butt AA, Shams S, Jabeen A, Al-Nuaimi AA, Krishnan JI, Malik AB, Saleem S, Abdulaziz MH, Seyam NI, Aziz K, Kandil D, Thomas AG, Nafady-Hego H, Lone MI, Al Ajmi J, Bhutta ZA, AlSulaiti N, Hussein WES, Semaan S, Al-Abdulla SA, Al-Kuwari MG, Abou-Samra AB. A prospective cluster randomized trial of an interventions bundle to reduce inappropriate antibiotic use for upper respiratory tract infections in the outpatient setting. BMC Infect Dis. 2025 Jul 1;25(1):818. doi: 10.1186/s12879-025-11210-z. PMID 40597774